CLINICAL TRIAL: NCT03658824
Title: Behavioural Activation for Bipolar Depression (BA-BD): A Case Series Evaluation
Brief Title: Behavioural Activation for Bipolar Depression: A Case Series
Acronym: BA-BD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Exeter (Other)
Collaborators: Devon Partnership NHS Trust (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 237525
Record Dates: First submitted 2018-07-26; First posted 2018-09-05 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Bipolar Depression
Keywords: Behavioural Activation; Bipolar Disorder; Bipolar Depression; Multiple Baseline; Case Series
MeSH Terms: conditions — Bipolar Disorder

STUDY DESIGN:
Intervention Model Description: This is a case series using a multiple baseline design whereby participants are randomly allocated to one of 6 durations of wait at baseline before commencing treatment.
Masking Description: It is not possible to blind the assessor to phase or baseline duration of participants in the case-series, as the length of time between assessments will reveal this. Nevertheless, the assessor and clients will be asked not to disclose which therapist is treating them. Use of self-report measures as the primary outcome measure is intended to minimise potential biases on the side of the researcher.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- 3 week wait (Other): Participant waits for 3 weeks after their baseline assessment before commencing therapy.
  Interventions: Other: Behavioural Activation (BA)
- 4 week wait (Other): Participant waits for 4 weeks after their baseline assessment before commencing therapy.
  Interventions: Other: Behavioural Activation (BA)
- 5 week wait (Other): Participant waits for 5 weeks after their baseline assessment before commencing therapy.
  Interventions: Other: Behavioural Activation (BA)
- 6 week wait (Other): Participant waits for 6 weeks after their baseline assessment before commencing therapy.
  Interventions: Other: Behavioural Activation (BA)
- 7 week wait (Other): Participant waits for 7 weeks after their baseline assessment before commencing therapy.
  Interventions: Other: Behavioural Activation (BA)
- 8 week wait (Other): Participant waits for 8 weeks after their baseline assessment before commencing therapy.
  Interventions: Other: Behavioural Activation (BA)

INTERVENTIONS:
Other: Behavioural Activation (BA) — BA is based on the assumption that depression may be precipitated and is maintained by a reduction in "healthy", adaptive behaviours and positive reinforcement of these, and an increase in avoidance behaviours. Together, these changes reduce the person's immediate distress, often at the expense of their medium and longer term goals. The therapy involves helping the individual to re-establish healthy patterns of activity, and replace avoidance behaviours with more adaptive behaviours that are constructive in the longer term.
  The intervention consists of up to 20 individual therapy sessions of Behavioural Activation, with one booster session three months after the end of therapy. Each session lasts approximately 50 minutes and this is supplemented by home practice between sessions.

SUMMARY:
Bipolar Disorders affect around 2% of the population. Most people with Bipolar experience depression; these periods can cause difficulties with relationships, work and daily life.

Psychological therapies for "unipolar" depression (for people who experience depression but never mania or hypomania) are widely available, but there is little research in to how effective these therapies are for people with Bipolar. Knowing this could give greater choice to people with Bipolar in terms of the therapy they have, and how easy it is to get within the NHS. One such therapy is called Behavioural Activation (BA). BA is an established therapy for people with unipolar depression. It helps people to re-establish healthier patterns of activity, but so far there is very little research into offering BA to people with BD.

The current research involves a small number of people with Bipolar Depression receiving BA to see if it seems sensible and worthwhile to them, and to help us to make any necessary improvements to the therapy. The study is taking place in Devon and is sponsored by the University of Exeter. 12 people that are currently experiencing Bipolar Depression who choose to take part will receive up to 20 individual therapy sessions of BA that has been adapted for Bipolar Depression (BA-BD), and will complete regular questionnaires and interviews. The results of this study will not give the final answer on how effective BA is for people with bipolar depression, but will help to plan for a larger study that can answer this question.

ELIGIBILITY:
Inclusion Criteria:

* scoring in the clinical range on a self-report measure of depression severity (the PHQ-9)
* meeting diagnostic criteria for depression based on a Structured Clinical Interview for Diagnosis (SCID-5)
* meeting diagnostic criteria for Bipolar I or II Disorder (SCID-5)
* participants will require working knowledge of written and spoken English, sufficient to be able to make use of therapy and to be able complete research assessments without the need of a translator.

Exclusion Criteria:

* current/past learning disability, organic brain change, substance dependence (drugs and alcohol) that would compromise ability to use therapy
* current marked risk to self (i.e. self-harm or suicide) that we deem could not be appropriately managed in the AccEPT clinic at the Mood Disorders Centre
* currently lacking capacity to give informed consent
* currently receiving other psychosocial therapy for depression or bipolar disorder
* presence of another area of difficulty that the therapist and client believe should be the primary focus of intervention (for example, Post-Traumatic Stress Disorder, psychosis).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
Minimally clinically significant improvement in depression symptoms for a majority of participants (>60%) | through study completion, an average of 7 months
  Participants' weekly completion of the Patient Health Questionnaire-9 (PHQ-9)
No significant adverse reaction for participants | through study completion, an average of 7 months
  Participant reports of adverse events elicited by researchers and therapists.
Qualitative feedback from participants | through study completion, an average of 7 months
  Written and verbal feedback of participants
Qualitative feedback from therapists | through study completion, an average of 7 months
  Feedback given in qualitative interviews with therapists
Therapy uptake rate | through study completion, an average of 7 months
  Number of participants randomised who attend at least 1 treatment session
Therapy completion rate | through study completion, an average of 7 months
  Proportion of participants that attend at least 8 treatment sessions

SECONDARY OUTCOMES:
Altman Self-Rating Mania Scale (ASRM) | 1 week
  5 item self-report measure of hypomania symptoms over the past week
Work and Social Adjustment Scale (WSAS) | 24 hours
  5 item self-report scale of functional impairment attributable to an identified problem
Structured Clinical Interview for Depression (SCID) | Six months
  Standardised interview to establish whether the participant meets research diagnostic criteria for lifetime Bipolar I or II Disorder, current depressive episode, and to establish whether they are experiencing current substance dependence
Hamilton Depression Scale (HAM-D) | 1 week
  17 item observer-rated scale measuring symptoms of depression over the past week
Brief Quality of Life in Bipolar Disorder (Brief QoLBD) | 1 week
  12 item self-report measure of disorder-specific quality of life
Bech-Rafaelsen Mania Scale | 1 week
  11 item observer-rated scale measuring the severity of manic states
Beck Depression Inventory (BDI) | 1 week
  21 item self-report measure of depressive symptoms and attitudes
General Anxiety Disorder Assessment - 7 (GAD7) | 2 weeks
  7 item self-report measure of anxiety symptoms
Behavioral Activation for Depression Scale (BADS) | 1 week
  25 item self-report measure of changes in activation and avoidance over the past week
Short Warwick-Edinburgh Mental Well-being Scale (SWEMWBS) | 2 weeks
  7-item self-report measure of wellbeing
Snaith-Hamilton Pleasure Scale (SHAPS) | 1 week
  14 item self-report measure of level of anhedonia
Positive and Negative Urgency Subscales of the UPPS-P Impulsive Behavior Scale | 6 months
  14 and 12 items respectively, these self-report scales measure tendency to respond impulsively to positive or negative feelings
Questions about Suffering, Struggling and Engagement in Valued Activities | 24 hours
  3 item self-report measure of core hypothesised process of change in behavioural activation, namely reduction in avoidance behaviours and increase in rewarding behaviours

CONTACTS AND LOCATIONS:
Overall Officials: Kim A Wright, PhD, Principal Investigator — University of Exeter
Locations (1):
- University of Exeter, Exeter, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
All data that underlie results in a publication.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Access will be possible from date of publication.
Access Criteria: The research database will be registered with the University of Exeter public access database. The dataset will be anonymous and will be registered with a metadata only record, allowing the research team to control access to the dataset, restricting it to appropriately qualified third parties.